CLINICAL TRIAL: NCT05598918
Title: Comparison of Early Passive and Active Mobilization Protocols in Flexor Tendon Repair Rehabilitation of the Hand, and Investigation of Factors Affecting the Results
Brief Title: Comparison of Early Passive and Active Mobilization Protocols in Flexor Tendon Repair Rehabilitation of the Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09.2021.118
Record Dates: First submitted 2022-08-03; First posted 2022-10-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-10

CONDITIONS: Tendon Injuries
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Intervention Model Description: The patients were divided into two groups as early active and passive mobilization groups. The angles of the dorsal orthoses of the active and passive groups were different. In the home exercise program in the active group, in addition to the exercises in the passive group, flexion was continued for 3-5 seconds at the end of passive flexion. The rehabilitation program was similar apart from these distinctions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients were randomized into two groups as active and passive rehabilitation groups by computer program. Patients, shear wave elastography practitioner and data evaluator were blinded to the treatment administered to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early passive mobilization (Experimental): ıt will begin to using an orthosis with 30* flexion of the wrist,70* flexion of metacarpophalangeal (MCP) joints,full extension of IF joints.Home exercises will be performed as passive flexion and active extension exercises with rubber band 10 times per hour on postoperative 3rd day for 3 weeks.Passive flexion and extension exercises will be performed ten times a day;four times a day on MCP+PIP+IF joints.3 weeks after repair and non-resistance active movement and tenodesis exercises will be started in presence of a physiotherapist.From the 6th week tendon gliding exercises and blocking exercises will be started.
  Interventions: Procedure: early passive mobilization
- early active mobilization (Experimental): ıt will begin to using an orthosis that positions wrist in neutral position,MCP joints 50*-70* flexion,IF joints in full extension.After flexion active extension exercises,full passive flexion of fingers with the other intact hand and then keeping fingers in flexion position for 3-5 sec for 3 weeks.Rehabilitation program applied from 3rd week is the same as the passive group:3 weeks after repair and non-resistance active movement and tenodesis exercises will be started in presence of a physiotherapist.From the 6th week tendon gliding exercises and blocking exercises will be started.
  Interventions: Procedure: early active mobilization

INTERVENTIONS:
Procedure: early active mobilization — In the active rehabilitation group, active extension and passive flexion of the metacarpophalangeal, proximal interphalangeal and distal interphalangeal joints were performed with kleinert splint at angles suitable for active mobilization group.Then, the patients were asked to passively flex the injured side with their healthy hand and hold it in the flexion position for 3-5 seconds.
  Arms: early active mobilization
Procedure: early passive mobilization — In the passive rehabilitation group, active extension and passive flexion of the metacarpophalangeal, proximal interphalangeal and distal interphalangeal joints were performed with kleinert splint at angles suitable for passive mobilization group.
  Arms: early passive mobilization

SUMMARY:
Many active and passive rehabilitation programs are applied in the rehabilitation processes after flexor tendon repair. There is no clear rehabilitation program accepted by the whole world. An accurate understanding of these injuries at the histological and biomechanical level is necessary to improve rehabilitation outcomes. Mechanical properties of tendons, such as their viscoelasticity, are affected by the increase in stiffness caused by the rupture, repair, and healing process. Previous studies have shown that the mechanical properties of a repaired tendon, such as stiffness, material properties and functionality of tendon tissue Shear-wave elastography can detect pathological changes in tendinopathy before they are visible on conventional Ultrasonography imaging. In addition, shear wave elastography allows the evaluation of quantitative measurements and is considered more objective because it provides reproducible results. Our aim in this study is to evaluate the changes in the mechanical properties of the hand flexor tendons repaired using shear wave elastography (SWE) during the rehabilitation process and natural process and their effect on functionality.

DETAILED DESCRIPTION:
Patients' affected tendons will be evaluated by shear wave elastography within 3 - 5 days after surgery. The tendons of the healthy hands of the patients will also be evaluated as the control group.

Afterwards, patients will be randomized into two groups by computer-assisted randomization.

Group 1: early passive mobilization Within 3 to 5 days following surgery, patients will begin using a dorsal forearm-based orthosis with 30* flexion of the wrist, 70* flexion of the metacarpophalangeal (MCP) joints, full extension of the interphalangeal (IF) joints. Home exercises will be performed as passive flexion and active extension exercises with rubber band 10 times per hour on the postoperative 3rd day for 3 weeks. Passive flexion and extension exercises will be performed ten times a day, four times a day, on the MCP + Proximal Interphalangeal (PIP) + IF joints. The bands will be removed at night and the fingers will be kept in full extension. In 3 weeks, the orthosis will be modified so that the wrist is in a neutral position and the MCP joints are extended a little more. Approximately 3 weeks after the repair, the dorsal orthosis will be removed during the exercises, and non-resistance active movement and tenodesis exercises will be started in the presence of a physiotherapist. From the 6th week, the dorsal orthosis will be worn only at night, tendon gliding exercises and blocking exercises will be started.

Group 2: early active mobilization Patients will begin to use a dorsal forearm-based orthosis that positions the wrist in a neutral position, metacarpophalangeal (MCP) joints 50* -70* flexion, IF joints in full extension within 3 to 5 days after surgery. After the flexion active extension exercises, full passive flexion of the fingers with the other intact hand and then gently keeping the fingers in the flexion position for 3-5 seconds when the contralateral hand is raised will be performed for 3 weeks, no force will be applied on the fingers. Passive flexion and extension exercises will be performed ten times a day, four times a day, on the MCP + PIP + IF joints. These exercises will be organized as a home exercise program. The patients will be evaluated by the physiotherapist and clinician once a week in the first two weeks of the exercises, and 3 days a week in the third week, in terms of monitoring the exercises, and the exercises will be shown again. The bands will be removed at night and the fingers will be kept in full extension. Approximately 3 weeks after the repair, the dorsal orthosis will be removed during the exercises, and the patients will be started with non-resistance active movement and tenodesis exercises in the form of a home exercise program 3 days a week with a physiotherapist on the remaining days. From the 6th week, the dorsal orthosis will be worn only at night, tendon gliding exercises and blocking exercises will be started.

Patients will be evaluated by an investigator blinded to the treatment groups at week 8 and week 12 using the following methods.

1. Tendon elasticity will be evaluated with shear wave elastography
2. Measurements of hand grip strength and pinch strength (only at 12 weeks) will be evaluated with a dynamometer device.
3. Duruoz Hand Index will be filled.
4. Total active movements of the fingers will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Forty patients aged 18-75 years who had flexor tendon injury and underwent primary surgical repair (within the first 10 days after injury) will be included in the study

Exclusion Criteria:

* Patients with a history of previous hand trauma, neurological or systemic disease affecting the hand, patients with a history of upper extremity surgery, concomitant extensor tendon injury, fracture and amputation will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level | T0 : Patients were evaluated on postoperative 5-7 days.
  Shear wave velocity, measured in metres per second, was recorded using shear wave elastography.
tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level | T1 : Patients were evaluated on postoperative 3 weeks.
  Shear wave velocity, measured in metres per second, was recorded using shear wave elastography.
tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level | T2 : Patients were evaluated on postoperative 8 weeks.
  Shear wave velocity, measured in metres per second, was recorded using shear wave elastography.
tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level tendon stiffness level | T3 : Patients were evaluated on postoperative 12 weeks.
  Shear wave velocity, measured in metres per second, was recorded using shear wave elastography.

SECONDARY OUTCOMES:
Handgrip strength | T0: Patients are evaluated on postoperative 12 weeks.
  The patient's handgrip strength, measured by JAMAR hand dynamometer, measured in Pounds.
Pinch grip strength | T0: Patients are evaluated on postoperative 12 weeks.
  The patient's pinch grip strength, measured by hydraulic pinch gauge, measured in Pounds.
Range of motion | T0: Patients are evaluated on postoperative 12 weeks.
  The range of motion of patient's fingers, measured by goniometer, measured in degrees.
Functionality | T0: Patients are evaluated on postoperative 12 weeks.
  Purdue peg board test, Nine hole test, measured in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, İ̇stanbul (asya), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirci M, Temiz Erguden FH, Sahbat Y, Bugdayci O, Baysal O, Sanal C. Active versus passive rehabilitation after flexor tendon repair: clinical outcomes and shear wave elastography monitoring in a randomized pilot study. Arch Orthop Trauma Surg. 2026 Jan 7;146(1):29. doi: 10.1007/s00402-025-06172-5. PMID 41498969